CLINICAL TRIAL: NCT02011295
Title: Bone Marrow Aspirate Concentrate Supplementation to Microfracture in the Treatment of Osteochondral Lesions of the Talus
Brief Title: Bone Marrow Aspirate Concentrate (BMAC) Supplementation for Osteochondral Lesions
Acronym: BMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00047251
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Osteochondral Lesions of Talus
Keywords: OLT; Surgical Intervention; BMAC
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microfracture (Other): Procedure/Surgery: ankle arthroscopy with debridement and microfracture of the OLT
  Interventions: Procedure: ankle arthroscopy with debridement and microfracture of the OLT
- microfracture + injection of autologous BMAC (Other): Procedure/Surgery: ankle arthroscopy with debridement and microfracture of the OLT plus injection of autologous Bone Marrow Aspirate Concentration
  Interventions: Procedure: ankle arthroscopy with debridement and microfracture of the OLT; Other: Bone Marrow Aspirate injection

INTERVENTIONS:
Procedure: ankle arthroscopy with debridement and microfracture of the OLT — ankle arthroscopy with debridement and microfracture of the OLT
Other: Bone Marrow Aspirate injection
  Arms: microfracture + injection of autologous BMAC

SUMMARY:
The purpose of this study is to determine the clinical efficacy of the application of bone marrow aspirate concentrate (BMAC) as a supplement to microfracture in the treatment of osteochondral lesions of the talus (OLTs).

DETAILED DESCRIPTION:
After appropriate patient identification and consent, patients will be asked to complete a 100 mm visual analog pain scale, a Foot and Ankle Disability Index questionnaire, a Short Form-36 questionnaire, and a Short Musculoskeletal Function Assessment questionnaire. They will then be randomized to one of two groups: (1) microfracture alone or (2) microfracture plus injection of autologous BMAC.

At the time of surgery, all patients will undergo standard ankle arthroscopy with debridement and microfracture of the OLT. If randomized to the microfracture alone group, no further intervention will take place. If randomized to the microfracture + BMAC group, then, while the surgeon is performing the ankle arthroscopy, the surgical assistant will perform the iliac crest bone marrow aspiration. The ipsilateral iliac crest will undergo sterile preparation and draped into the surgical field. The iliac crest aspiration site will be injected with 2cc of 1% lidocaine for postoperative pain control. Through an approximate 4mm incision, approximately 2 cm posterior to the patient's ipsilateral anterior superior iliac spine, a Jamshidi® type trocar/cannula system will be placed through the incision and the medial and lateral borders of the pelvic brim will be palpated. Once centered, the needle will be malleted into the pelvis between the inner and outer tables to a depth of 2-3 cm. The sharp trocar will be switched for the blunt trocar and introduced another 2-3cm. The blunt trocar is used to prevent penetration of the cannula through the inner table cortex. Next, 60cc of iliac crest bone marrow will be aspirated. The needle will be withdrawn and the incision is closed with one 3-0 nylon suture. The iliac crest bone marrow aspirate is then passed through a filter to remove any bone spicules and then centrifuged using the Harvest SmartPReP 2 BMAC system (http://www.harvesttech.com). This device is approved for intra-operative point-of-care use for concentrating iliac crest bone marrow. Its use is approved at Duke. The process takes approximately 15 minutes and will be occurring simultaneous to the ankle arthroscopy, debridement, and microfracture of the OLT. Concentration of 60cc of iliac crest bone marrow aspirate typically yields 6-7cc of BMAC. Therefore, to provide a standard amount of BMAC across all cases, 5cc of the BMAC will be injected into the ankle joint through the arthroscopy incision prior to closure.

All patients will be placed in a postoperative splint and remain non-weightbearing for six weeks as a standard protocol for microfracture of OLTs. They will return for the first postoperative visit 2-3 weeks after the surgery and the sutures will be removed.

Additional post-surgical routine follow-up occurs at 3 months, 6 months, 1 year, and 2 years. These standard time-points will occur for all patients enrolled in this study. At each time-point, patients will be asked to complete a 100 mm visual analog pain scale, a Foot and Ankle Disability Index questionnaire, a Short Form-36 questionnaire, and a Short Musculoskeletal Function Assessment questionnaire. At the one-year time-point, patients will be scheduled for a repeat MRI.

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* has an OLT that has not had previous surgical treatment

Exclusion Criteria:

* OLT greater than 1.5cm in diameter (these require more extensive treatment)
* more than one OLT
* radiographic evidence of widespread ankle joint arthritis
* any systemic inflammatory disease
* any ankle deformity

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Pain Assessment | pre-operative up to 2yrs post surgery
  Visual Analog Scale (VAS)
Change in Functional Assessment | pre-operative to 2yrs post surgery
  Foot and Ankle Disability Index

SECONDARY OUTCOMES:
Change in Functional Assessment | pre-operative through 2yrs post surgery
  Short Form 36 (SF36)
Change in Functional Assessment | pre-operative through 2yrs post surgery
  Short Musculoskeletal Function Assessment (SMFA)
MRI Assessment | 1 year post surgical intervention
  Measurement of lesion and bone marrow edema size

CONTACTS AND LOCATIONS:
Overall Officials: Samuel B Adams, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States